CLINICAL TRIAL: NCT02472678
Title: Web-based Tailored Information and Support for Patients With a Neuroendocrine Tumor
Acronym: WIN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20150501
Record Dates: First submitted 2015-01-06; First posted 2015-06-16 (Estimated); Last update posted 2024-05-06 (Actual); Status verified 2024-05

CONDITIONS: Neuroendocrine Tumor
MeSH Terms: conditions — Neuroendocrine Tumors | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard care (Other): The control group will receive standard care.
  Interventions: Other: Standard care
- Experimental group (Experimental): In addition to standard care, the experimental group will be given access to the web-based tailored information and support system (with a username/password)
  Interventions: Other: Web-based tailored information and support system

INTERVENTIONS:
Other: Web-based tailored information and support system — Access to the web-based tailored information and support system (with a username/password)
  Arms: Experimental group
Other: Standard care — The control group will receive standard care.
  Arms: Standard care

SUMMARY:
Patients with a neuroendocrine tumor (NET) frequently suffer from physical as well as psychosocial complaints. Patients may experience various symptoms from tumor burden and secreted hormones by the tumor. They also can have complaints due to their anti-cancer treatment and accompanying side effects.

Adequate information is an essential aspect of supportive care. Patients need for information and care remain frequently unnoticed. The aim of the current study is to test the effectiveness of a web-based tailored information and support system to support patients' information and care needs. Key features of this website are patient self-screening of physical and psychosocial problems, tailored patient education on reported problems and self-referral to professional health care. The investigators expect that the website is a highly suitable medium to provide tailored information and support.

DETAILED DESCRIPTION:
Rationale: Patients with a neuroendocrine tumor (NET) frequently suffer from physical as well as psychosocial complaints. Patients may experience various symptoms from tumor burden and secreted hormones by the tumor. They also can have complaints due to their anti-cancer treatment and accompanying side effects.

Adequate information is an essential aspect of supportive care. Patients need for information and care remain frequently unnoticed. The aim of the current study is to test the effectiveness of a web-based tailored information and support system to support patients' information and care needs. Key features of this website are patient self-screening of physical and psychosocial problems, tailored patient education on reported problems and self-referral to professional health care. The invetigators expect that the website is a highly suitable medium to provide tailored information and support.

Objective: This study has a combined objective to investigate whether a web-based tailored information and support system reduces distress, as determined by a decrease in value of the distress thermometer, and/or improves patients' perception and satisfaction of received information, as determined by an improved score at the EORTC QLQ-INFO 25 questionnaire, as compared to patients who receive standard care.

Secondary aims are improvement in quality of life as determined by the cancer-specific EORTC QLQ-C30 and the NET-specific EORTC QLQ-GINET21, empowerment at end of study (subscales of the Construct Empowering Outcomes questionnaire) and to investigate patients' opinion about and use of the web-based tailored information and support system (with a self-constructed questionnaire; based on constructs of the Technology Acceptance Model (TAM) questionnaire and two self-constructed questions).

Study design: The present study is a single center randomized, prospective, intervention study on the efficacy of a tailored web-based information and support system in NET patients. After randomization and stratification - based on the time from diagnosis till inclusion- the control group receives standard care and the experimental group receives the standard care complemented with use of the web-based tailored information and support system for 12 weeks.

Patients will be asked to fill out questionnaires at baseline and after 12 weeks.

Patients in the intervention group are asked to fill out an extra questionnaire about use of the web-based tailored information and support system.

Study population: Diagnosed NET patients who are under treatment at the Department of Medical Oncology in the University Medical Center Groningen will be invited to participate in the study. The investigators will stratify for newly diagnosed patients (diagnosed within six months before inclusion) and patients diagnosed more than 6 months before inclusion

ELIGIBILITY:
Inclusion Criteria:

* Adult NET patients (aged ≥ 18 years of age) with any tumor site and disease stage.
* Ability to comprehend Dutch (both reading and writing).
* Informed consent provided

Exclusion Criteria:

* Estimated life expectancy less than 3 months.
* Patients who have a history of another primary malignancy, except for radical and adequately treated malignancies from which the patient has been disease free for ≥ 3 years
* Patients who participated in the WIN-pilot study.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2015-05; Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
A composite outcome of difference in distress and the mean improvement of the global score of the EORTC QLQ-INFO 25 | 12 weeks
  The primary endpoint is a composite of the difference in distress measured by the distress thermometer and the mean improvement of the global score of the EORTC QLQ-INFO 25 at end of study between the control group and the intervention group.

SECONDARY OUTCOMES:
change in quality of life, | 12 weeks
  change in quality of life as determined by the cancer-specific EORTC QLQ-C30, and the EORTC QLQ-GINET21,
Empowerment at end of study | 12 weeks
  empowerment at end of study (subscales of the Construct Empowering Outcomes questionnaire)
Information about patients' opinion and use of the web-based tailored information and support system | 12 weeks
  investigation of patients' opinion about and use of the web-based tailored information and support system (with a self-constructed questionnaire; based on constructs of the Technology Acceptance Model (TAM) questionnaire and two self-constructed questions

CONTACTS AND LOCATIONS:
Overall Officials: A. M.E. Walenkamp, MD, PhD, Principal Investigator — University Medical Center Groningen
Locations (1):
- University Medical Center Groningen, Groningen, Netherlands

REFERENCES:
- [Derived] de Hosson LD, Bouma G, Stelwagen J, van Essen H, de Bock GH, de Groot DJA, de Vries EGE, Walenkamp AME. Web-based personalised information and support for patients with a neuroendocrine tumour: randomised controlled trial. Orphanet J Rare Dis. 2019 Feb 28;14(1):60. doi: 10.1186/s13023-019-1035-3. PMID 30819238